CLINICAL TRIAL: NCT07295743
Title: The Effect of Implant Prosthesis Emergence Angle on Peri-Implant Health and Disease
Brief Title: Effect of Emergence Angle on Peri-implant Status
Acronym: EEAPS
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-DH-TS-04
Record Dates: First submitted 2025-11-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Peri-implant Health
Keywords: Dental implants; Emergence angle; Peri-implantitis; Peri-implant tissue
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peri-implantitis: Peri-implantitis patients are those who have developed inflammation around a dental implant, leading to the loss of supporting bone and the presence of pockets of infection.
  Interventions: Other: emergence profile
- Peri-implant mucositis: Peri-implant mucositis refers to a reversible inflammatory condition affecting the soft tissues surrounding a dental implant, characterized by redness, swelling, and bleeding on probing, without any bone loss.
  Interventions: Other: emergence profile
- Peri-implant health: Peri-implant health refers to the condition where the tissues surrounding a dental implant are free from inflammation, with no signs of redness, swelling, bleeding on probing, or bone loss, indicating a stable and healthy implant environment.
  Interventions: Other: emergence profile

INTERVENTIONS:
Other: emergence profile — The emergence angles of the implants were measured on panoramic radiographs.

SUMMARY:
The study was conducted at the Division of Periodontology, Bolu Abant İzzet Baysal University Faculty of Dentistry. Participants were systemically healthy individuals aged 18 to 70 who had received dental implant prostheses within the past five years and had high-quality panoramic radiographs. The peri-implant status of the subjects was evaluated using various indices and radiographic analyses in accordance with Chicago's Classification of Periodontal and Peri-Implant Diseases and Conditions. Additionally, measurements of gingival thickness, gingival phenotype, keratinized gingival width, and emergence angle were performed.

DETAILED DESCRIPTION:
Patient histories were collected from those who met the study criteria, and panoramic radiographs were taken. A total of 310 implants were initially assessed, and 192 implants were selected for inclusion in the study. All implant patients underwent an evaluation of plaque index , gingival index, bleeding on probing , pocket depth, clinical attachment level, and gingival recession. The peri-implant condition was determined using these indices and radiographs, in accordance with the guidelines from the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions and the 2023 European Federation of Periodontology. Patients were categorized into three groups: peri-implantitis (64), peri-implant health (64), and peri-implant mucositis (64). Additionally, gingival thickness (GT), keratinized gingival width (KGW), and gingival phenotype (GP) around the implants were measured, and the emergence angle (EA) of the implants was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals or individuals with controlled medical conditions
* Availability of high-quality panoramic radiographs that could be accurately measured after fabrication of the dental implant prosthesis
* Implants placed no more than five years prior to evaluation

Exclusion Criteria:

* Individuals with uncontrolled systemic diseases
* Presence of habitual bruxism
* Current smokers
* Pregnant or breastfeeding individuals
* Use of anti-inflammatory or immunosuppressive medications affecting the mucosa or bone
* Individuals who had received treatment for peri-implant disease after implant placement
* Development of peri-implantitis due to residual cement or prosthesis design, or improperly positioned implants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have received implants
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Emergence angle | Baseline
  EA was determined by measuring the angle formed between the long axis of the implant and a tangent line drawn to the restoration. A line was initially drawn along the long axis of the implant at its outside collar. Subsequently, a second line, tangent to the restoration, was drawn from the platform. The angle at which the junction occurred was recorded as the EA .

SECONDARY OUTCOMES:
periodontal pocket depth | Baseline
  The periodontal pocket depth is the measurement of the distance between the gingival margin and the most coronal region of the junctional epithelium.
bleeding on probing | Baseline
  The bleeding on probing index was established as the occurrence of bleeding in the sulcus, thirty seconds after measuring the depth of the periodontal pockets in all dental implant.
plaque index | Baseline
  an index for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin. 0 is minimum and 3 is maximum. The situation worsens as the score increases.
gingival index | Baseline
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding. 0 is minimum and 3 is maximum.
clinical attachment level | Baseline
  The peri-implant clinical attachment level is determined by measuring the distance from the implant margin to the base of the mucosal sulcus using a Williams periodontal probe.
Gingival recession | Baseline
  Gingival recession is the measured distance between the enamel-cementum and the gingival margin. Assessment was performed using a Williams periodontal probe.
gingival thickness | Baseline
  GT was measured by inserting a number eight canal file from the buccal side of the implant until it reached the alveolar bone and then securing it with a stopper to determine the distance.
keratinized tissue width | Baseline
  The width of the keratinized gingiva was measured via a periodontal probe from the mucogingival margin to the gingival margin.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Şahin, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Dentistry Faculty, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided